CLINICAL TRIAL: NCT03401515
Title: Using Propranolol in Traumatic Brain Injury to Reduce Sympathetic Storm Phenomenon: A Prospective Randomized Clinical Trial Injury to Reduce Sympathetic Storm Phenomenon: A Prospective Randomized Clinical Trial
Brief Title: Using Propranolol in Traumatic Brain Injury to Reduce Sympathetic Storm Phenomenon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Lecturer of anesthesia,intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1345 AUS
Record Dates: First submitted 2017-11-21; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propranolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Adminstration of propranolol hydrochloride ( 1 MG /ml) 1 mg every 6 hrs .
  Interventions: Drug: Propranolol Hydrochloride 1 MG/ML
- Control (Placebo Comparator): Adminstration of normal saline 1 mg every 6 hrs
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Propranolol Hydrochloride 1 MG/ML — Propranolol 1 mg every 6 hrs in the first 24 hrs after isolated blunt traumatic brain injury
  Arms: Intervention
Other: Normal saline — Normal Saline 1 ml every 6 hrs
  Arms: Control

SUMMARY:
Traumatic Brain Injury (TBI) is one of the leading causes of death. Severe TBT is correlated with an exaggerated stress response due to plasma catecholamine levels known as sympathetic storming. It is also autonomic dysfunction syndrome. This phenomenon is also associated with brain tumors, severe hydrocephalus and subarachnoid hemorrhage. Patients are presented by tachycardia, tachypnea hypertension, diaphoresis, dystonia, hyperthermia, and dilated pupils with elevated levels of plasma catecholamine and blood glucose .

DETAILED DESCRIPTION:
The sympathetic storming events can be triggered by suctioning, repositioning, or environmental stimuli. To differentiate sympathetic storming from similar conditions, symptoms and signs have to occur in TBI patients a minimum of 1 cycle per day for 3 consecutive days (body temperature of 38.5 °C or more, heart rate at least 120 beat / min, systolic blood pressure > 140 mmHg, respiratory rate > 20 breaths / min, in presence of dystonia, diaphoresis, agitation and laboratory investigations confirm elevated serum catecholamines. Beta blockers has a cardio protective effect via lowering heart rate, stroke volume and mean arterial blood pressure which limits myocardial O2 consumptions and guards against myocardial infarction. They also have neuron protective effects via reducing cerebral blood flow thus lowering O2 and glucose consumption as cerebral metabolism is reduced. Propranolol a nonselective B receptor antagonists works on β1 receptors in brain, heart, and kidney and β 2 receptors in lungs, liver, skeletal muscles, eye and arterioles.We suppose that using Beta - adrenergic receptor blockers as propranolol blunts the sympathetic storming phenomenon as it is a nonselective β inhibitor and has a lipophilic property which enables it to penetrate blood brain barrier.

ELIGIBILITY:
Inclusion criteria:

* Patients with isolated blunt TBI
* From 18 to 60 years old both sex
* Not in need of mechanical ventilation
* GCS on admission between 9 and 12
* Rotterdam CT score from 2-4.
* Normal Procalcitonin test to exclude infection.

Exclusion criteria:

* Preexisting heart disease
* Myocardial injury
* Craniotomy
* Preexisting cerebral dysfunction
* Spinal cord injury
* Diabetes mellitus
* Severe liver or kidney disease
* Patients with sepsis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
catecholamine level | 7 days
  Norepinephrine plasma levels in pg./ml

SECONDARY OUTCOMES:
Temperature | 7 days
  Temperature in °C